CLINICAL TRIAL: NCT04695132
Title: Illness Management and Recovery- en behandlingsutvärdering Inom rättspsykiatrin.
Brief Title: Illness Management and Recovery- a Cluster Randomized Controlled Trial Within a Forensic Mental Inpatient Setting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Karolinska Institutet (Other)
Collaborators: Dalarna County Council, Sweden (Other)
Responsible Party: Principal Investigator, Knut Sturidsson, Lecturer/PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20211805
Record Dates: First submitted 2020-11-23; First posted 2021-01-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Psychotic Disorders; Forensic Psychology; Forensic Nursing; Antisocial Personality Disorder; Substance Use Disorders
MeSH Terms: conditions — Psychotic Disorders; Antisocial Personality Disorder; Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to one of two arms: Active treatment arm (recipients of Illness Management and Recovery) and Control condition (TAU). Participants in the Control condition will be offered Illness Management and Recovery after study completion, conditional on them still being treated at the forensic inpatient treatment sites that are part of the study. Participants will be recruited in clusters (consisting of wards at inpatient treatment sites) and enrollment of new clusters will take place continually during data collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Illness Management and Recovery treatment programme (intervention group) (Experimental): These patients receive the Illness Management and Recovery treatment. Treatment takes place during 2 Group sessions and 1 individual session per week.
  Interventions: Behavioral: Illness Management and Recovery treatment programme
- Treatment as usual (control group) (No Intervention): These patients receive treatment as usual consisting of the standard treatment given at the respective inpatient forensic mental health facility where they are admitted.

INTERVENTIONS:
Behavioral: Illness Management and Recovery treatment programme — The Illness Management and Recovery treatment programme is a psychosocial treatment aimed at attaining illness management skills and promoting a sense of personal recovery amongst patients with serious mental illness. The original treatment protocol has been translated to Swedish and adapted to a forensic mental health setting. The treatment consists of ten chapters containing information and practical exercises relating to topics relevant for mental health and mental health recovery. These topics include medication use, stress reduction, problem solving, recovery goals and navigating the forensic mental health system. Participants are assigned practical homework and tasks to be completed outside of treatment sessions. Group sessions are conducted to present and discuss treatment material. Individual sessions are used to rehearse treatment content, personalize the treatment and review progress in achieving tasks agreed upon in the group setting.
  Arms: Illness Management and Recovery treatment programme (intervention group)

SUMMARY:
The purpose of the study is to investigate the effects of a psychoeducational intervention program, Illness Management and Recovery (henceforth abbreviated as IMR), when administered to inpatient forensic mental health patients. IMR is a treatment program that can be administered in both a group and an individual format. It is designed for persons suffering from severe mental health problems and has two principal aims: 1. promoting participants´ capacity to manage and alleviate symptoms and functional impairment and 2. helping participants in formulating and attaining subjectively meaningful recovery goals. Forensic mental health inpatients receiving this treatment will be compared to patients who receive treatment as usual on a variety of outcome measures, such as clinician and self-rated levels of symptoms, function and perceived levels of hope. Furthermore, clinicians' experiences of working with the intervention will be investigated using a structured questionnaire regarding implementation processes and through an interview protocol.

The study has 3 objectives:

1. Investigating the effects of the treatment on the chosen outcome measures.
2. Investigating the effects of potential moderators on treatment outcome. These moderators include: pre-treatment functional status measured by self and informant report, neuropsychological performance and pre-admission indicators of presence of criminogenic risk factors and everyday functioning.
3. Investigating the experiences of staff working with the intervention, through the lense of Normalization Process Theory.

DETAILED DESCRIPTION:
The plan is to conduct the study through a cluster-randomized approach. Recruitment will take place amongst inpatients in the Swedish forensic mental health services. The clusters of patients randomized to the two study conditions will in effect be inpatient forensic mental health wards at Swedish forensic facilities. Enrolment and randomizing of clusters will take place stepwise during the duration of the study. Inpatient wards at participating sites will be randomized to either the control or the active condition and patients at these wards will be asked to give informed consent before participating in the study. After training, the staff at these wards will administer IMR to patients during two group sessions and one individual session a week. The IMR treatment administered consist of 10 chapters containing information and exercises pertaining to subjects relevant to mental health and recovery, such as medication use, social support, problem solving, etc. Translation of the original IMR-manual into Swedish and adaptions to the forensic mental health setting was done with permission from the original developers and authors of the treatment protocol. Study participants at control wards will receive treatment as usual. Data collection takes place at four times during the study (before start of treatment, four months into treatment, post treatment and during a three month follow-up). During data collection, participants fill in self-report measurements of symptom levels, functional impairment and perceived hope. Clinicians with good knowledge of participants also complete informant questionnaires on perceived levels of patient symptoms and functioning. During the data collection that takes place before treatment, participants also complete a neuropsychological test ("Zoo park" from the Behavioral assessment of dysexecutive syndrome, BADS). Anamnestic data pertaining to the pre-admission functioning and criminal history of the patients in the active condition will also be collected from the patient files. The data collection mentioned in the previous two sentences will be done to investigate potential moderators of treatment outcomes.

The outcome measures used in the study are WHODAS 2.0 (World Health Organization Disability Schedule 2.0 self-report and informant versions), IMRs (Illness management and Recovery treatment scale, self-report and informant versions), HoNOS-S (Health of Nation Outcome Scale-Secure version) and ASHS (Adult State Hope Scale). During the data collection four months into treatment, only IMRs and ASHS is completed, whereas all outcome scales are completed during the other data collection points. During the data collection post-treatment, treatment participants also complete CSQ-8 (Client Satisfaction Questionnaire-8).

The experiences of the staff administrating the treatment also will be investigated, with the purpose of exploring the process of implementing the intervention in this setting. This will be done using the Swedish version of the NoMAD-questionnaire (Normalization Process Theory Measure), which is a tool developed to operationalize the theoretical framework of Normalization Process Theory. The staff will complete this questionnaire after receiving training in the intervention, three months after treatment commencement and during a follow-up a year after treatment commencement. During the latter two of these data collection points staff will also be interviewed in a semi-structured fashion, using the questions in the NoMAD-questionnaire as a starting point for collection of more in depth qualitative data on the implementation of IMR. The part of the study pertaining to staff experiences of working with IMR are exploratory in character and we do not consider NoMAD to be a measure of treatment outcome.

As mentioned above, certain anamnestic data and neuropsychological performance (measured by the Zoo-map subtest), will be collected and analyzed as potential moderators of treatment outcome. The pre-treatment self and informant-report of everyday functioning (measured by WHODAS 2.0) will also be analyzed as a potential moderator of treatment effects on the other outcome measures. Of special interest in this regard will be discrepancies between the participants´ self reported functional status (assessed by WHODAS 2.0 self report) and other measures of functional status (informant version of WHODAS 2.0, performance on the Zoo map-test and anamnestic indicators of functioning). This interest is motivated by previous research indicating that overestimation of own abilities play a part in predicting outcomes for schizophrenia spectrum patients.

ELIGIBILITY:
Inclusion Criteria:

* Recipient of court mandated forensic mental health care following conviction of crime and diagnosis of serious mental illness
* Deemed capable of giving informed consent to research by treating medical staff

Exclusion Criteria:

* Recipient of treatment for other reason than court mandated care (e.g., recipients of prison sentences receiving temporary mental health treatment, patients receiving compulsory mental care without previous conviction of crime)
* Deemed uncapable or unwilling to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Health of Nation Outcome Scale-Secure version (HoNOS-S) (change from baseline levels to post treatment, estimated approximately 9 months after baseline). | This comparison will be made between HoNOS ratings in treatment and control group taken before treatment commencement and directly following treatment completion (estimated 9 months in between)
  An informant rating scale answered by the participants treating psychiatrists. The scale provides information on informant assessment of the participants level of symptom burden, functioning and the perceived need of special security measures in the care of the patient. The scale consists of a total of 19 items, 12 pertaining to clinical factors regarding perceived symptom burden and level of functioning and 7 pertaining to the perceived necessity of security arrangements associated with the care of the individual participant/patient.
World Health Organizations Disability Assessment Schedule 2.0 36-item version, interview administered. (change from baseline levels to post treatment estimated 9 months after baseline). | This comparison will be made between WHODAS ratings in treatment and control group taken before treatment commencement and directly following treatment completion (estimated 9 months in between)
  An interviewed schedule designed to measure the respondents health and level of disability. Measures this in six subdomains (cognition, mobility, personal care, relations, daily activities and participation). Research participants are interviewed with this assessment schedule.

SECONDARY OUTCOMES:
Illness Management and Recovery Scale-Self report version (change from baseline to measure taken 4 months after treatment start) | Control and active group´s change scores between baseline measure and 4-months after treatment commencement will be compared.
  A questionnaire designed to measure progress towards the goals stipulated in Illness Management and Recovery. The questionnaire contains 15 items answered on a scale from 1-5. Items include queries on the respondents self-assessment of own level of knowledge regarding mental illness, their access to social support and the presence of a clear plan for illness management.
Illness Management and Recovery Scale-Self report version (change from baseline to post-treatment completion, estimated 9 months in between). | Control and active group´s change scores between baseline measure and treatment completion (estimated to 9 months in between) will be compared.
  A questionnaire designed to measure progress towards the goals stipulated in Illness Management and Recovery. The questionnaire contains 15 items answered on a scale from 1-5. Items include queries on the respondents self-assessment of own level of knowledge regarding mental illness, their access to social support and the presence of a clear plan for illness management.
Illness Management and Recovery Scale-Self report version (change from baseline to 3 months follow up after treatment completion, estimated time 12 months in between). | Control and active group´s change scores between baseline measure and follow up 3 months after treatment completion (estimated time 12-months between the measures) will be compared.
  A questionnaire designed to measure progress towards the goals stipulated in Illness Management and Recovery. The questionnaire contains 15 items answered on a scale from 1-5. Items include queries on the respondents self-assessment of own level of knowledge regarding mental illness, their access to social support and the presence of a clear plan for illness management.
Illness Management and Recovery Scale- Clinician administered version (change from baseline to follow up 4 months after treatment start) | Control and active group´s change scores between baseline measure and 4-months after treatment commencement will be compared.
  A questionnaire designed to measure progress towards the goals stipulated in Illness Management and Recovery. The questionnaire contains 15 items answered on a scale from 1-5. This version is administered to a clinician with good knowledge of the research participant. Items include queries on the respondents assessment of the participants level of knowledge regarding mental illness, their access to social support and the presence of a clear plan for illness management.
Illness Management and Recovery Scale- Clinician administered version (change from baseline to post-treatment completion, estimated 9 months in between). | Control and active group´s change scores between baseline measure and treatment completion (estimated to 9 months in between) will be compared.
  A questionnaire designed to measure progress towards the goals stipulated in Illness Management and Recovery. The questionnaire contains 15 items answered on a scale from 1-5. This version is administered to a clinician with good knowledge of the research participant. Items include queries on the respondents assessment of the participants level of knowledge regarding mental illness, their access to social support and the presence of a clear plan for illness management.
Illness Management and Recovery Scale- Clinician administered version (change from baseline to 3 months follow up after treatment completion, estimated time 12 months in between). | Control and active group´s change scores between baseline measure and follow up 3 months after treatment completion (estimated time 12-months between the measures) will be compared.
  A questionnaire designed to measure progress towards the goals stipulated in Illness Management and Recovery. The questionnaire contains 15 items answered on a scale from 1-5. This version is administered to a clinician with good knowledge of the research participant. Items include queries on the respondents assessment of the participants level of knowledge regarding mental illness, their access to social support and the presence of a clear plan for illness management.
World Health Organizations Disability Assessment Schedule 2.0 36-item version, proxy administered, change between baseline and measure taken after treatment completion (estimated 9 months in between the two measures) | Change scores on the proxy version of WHODAS from baseline measure to a measure taken after treatment completion (estimated 9 months in between) will be compared between active and control group.
  A proxy administered version of WHODAS designed with the same purpose as the interview version: to assess a persons health and level of disability, in this version by posing questions regarding this to a proxy informant. Measures this in six subdomains (cognition, mobility, personal care, relations, daily activities and participation). Care staff with good knowledge of research participants answer this questionnaire.
World Health Organizations Disability Assessment Schedule 2.0 36-item version, proxy administered (change from baseline to 3 months follow up after treatment completion, estimated time 12 months in between). | This comparison will be made between scores for control and active group on proxy measures of WHODAS at baseline and a 3 months follow up after completion (i.e. approx. 12 months after baseline measure at treatment start)
  A proxy administered version of WHODAS designed with the same purpose as the interview version: to assess a persons health and level of disability, in this version by posing questions regarding this to a proxy informant. Measures this in six subdomains (cognition, mobility, personal care, relations, daily activities and participation). Care staff with good knowledge of research participants answer this questionnaire.
Adult State Hope Scale (ASHS) (change from baseline to measure taken 4 months after treatment start) | Control and active group´s change scores between baseline measure and 4-months after treatment commencement will be compared.
  A self-rating instrument designed to measure the respondents level of hope by 6-items answered on a 8-point scale.
Adult State Hope Scale (ASHS) (change from baseline to post-treatment completion, estimated 9 months in between). | Control and active group´s change scores between baseline measure and treatment completion (estimated to 9 months in between) will be compared.
  A self-rating instrument designed to measure the respondents level of hope by 6-items answered on a 8-point scale.
Adult State Hope Scale (ASHS) (change from baseline to 3 months follow up after treatment completion, estimated time 12 months in between). | Control and active group´s change scores between baseline measure and follow up 3 months after treatment completion (estimated time 12-months between the measures) will be compared.
  A self-rating instrument designed to measure the respondents level of hope by 6-items answered on a 8-point scale.
World Health Organizations Disability Assessment Schedule 2.0 36-item version, interview administered. (change from baseline to 3 months follow up after treatment completion, estimated time 12 months in between). | This comparison will be made between WHODAS ratings in treatment and control group taken at baseline and a 3 months follow up after treatment completion (i.e. approx. 12 months after treatment start)
  An interviewed schedule designed to measure the respondents health and level of disability. Measures this in six subdomains (cognition, mobility, personal care, relations, daily activities and participation). Research participants are interviewed with this assessment schedule.
Health of Nation Outcome Scale-Secure version (HoNOS-S) (change from baseline to 3 months follow up after treatment completion, estimated time 12 months in between). | This comparison will be made between HONOS ratings in treatment and control group taken at baseline and a 3 months follow up after treatment completion (i.e. approx. 12 months after treatment start)
  An informant rating scale answered by the participants treating psychiatrists. The scale provides information on informant assessment of the participants level of symptom burden, functioning and the perceived need of special security measures in the care of the patient. The scale consists of a total of 19 items, 12 pertaining to clinical factors regarding perceived symptom burden and level of functioning and 7 pertaining to the perceived necessity of security arrangements associated with the care of the individual participant/patient.

OTHER OUTCOMES:
Normalization Process Theory Measure Swedish version (S-NoMAD) (12 months after treatment start) | This measurement takes place 12 months after treatment commencement.
  S-NoMAD is a measure developed to measure different aspects of implementation processes within the healthcare sector according to how those processes are conceptualised within Normalization Process Theory. The scale covers the four core constructs of implementation work postulated within Normalization Process Theory (Coherence, Cognitive Participation, Collective Action, Reflexive Monitoring). This measure is administered to staff at wards where IMR is implemented. The purpose of this is to explore staff experiences of working with IMR. During this assessment point, participants also complete a semi-structured group interview based on a qualitative expansion of the S-NoMAD.
Normalization Process Theory Measure Swedish version (S-NoMAD) (before treatment start) | This measure is answered by staff administrating treatment, after of preparatory training approximately 2 weeks before treatment commencement.
  S-NoMAD is a measure developed to measure different aspects of implementation processes within the healthcare sector according to how those processes are conceptualised within Normalization Process Theory. The scale covers the four core constructs of implementation work postulated within Normalization Process Theory (Coherence, Cognitive Participation, Collective Action, Reflexive Monitoring). This measure is administered to staff at wards where IMR is implemented. The purpose of this is to explore staff experiences of working with IMR.
Normalization Process Theory Measure Swedish version (S-NoMAD) (3-months after treatment start). | This measurement takes place 3 months after treatment commencement.
  S-NoMAD is a measure developed to measure different aspects of implementation processes within the healthcare sector according to how those processes are conceptualised within Normalization Process Theory. The scale covers the four core constructs of implementation work postulated within Normalization Process Theory (Coherence, Cognitive Participation, Collective Action, Reflexive Monitoring). This measure is administered to staff at wards where IMR is implemented. The purpose of this is to explore staff experiences of working with IMR. During this assessment point, participants also complete a semi-structured group interview based on a qualitative expansion of the S-NoMAD.
Illness Management and Recovery Treatment Integrity Scale (IT-IS) ( approx. 3-months after treatment start) | The first audio recording of an IMR session in the active group, is scheduled to take place approximately 3 months after the treatment start.
  IT-IS is an instrument developed to assess a healthcare professionals fidelity to the treatment manual whilst administering IMR. It contains 16 items (13 mandatory items, 3 optional). It is designed to be scored by an IMR-proficient clinician whilst observing a session. In this study, this instrument is used to assess the quality of the treatment delivered to participants in the treatment condition. Audio recordings are made of 2 treatment sessions per cluster within the active treatment group and are used to score treatment fidelity with IT-IS. The scoring of IT-IS is made by the research team.
Illness Management and Recovery Treatment Integrity Scale (IT-IS) (approx. 5-months after treatment start). | The second audio recording of an IMR session in the active group, is scheduled to take place approximately 5 months after the treatment start.
  IT-IS is an instrument developed to assess a healthcare professionals fidelity to the treatment manual whilst administering IMR. It contains 16 items (13 mandatory items, 3 optional). It is designed to be scored by an IMR-proficient clinician whilst observing a session. In this study, this instrument is used to assess the quality of the treatment delivered to participants in the treatment condition. Audio recordings are made of 2 treatment sessions per cluster within the active treatment group and are used to score treatment fidelity with IT-IS. The scoring of IT-IS is made by the research team.
Client Satisfaction Questionnaire-8 (CSQ-8) | This questionnaire is answered by research participants in the active condition after treatment completion (estimated 9-months after treatment start).
  CSQ-8 is a self-report questionnaire used to assess a respondents level of satisfaction with a treatment programme. The questionnaire contains 8 questions answered on a scale from 1-4. A brief semi-structured interview is also conducted with the respondent.

CONTACTS AND LOCATIONS:
Overall Officials: Knut Sturidsson, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Rättspsykiatriska kliniken i Sala, Sala, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Andersson P, Tistad M, Eriksson A, Enebrink P, Sturidsson K. Implementation and evaluation of Illness Management and Recovery (IMR) in mandated forensic psychiatric care - Study protocol for a multicenter cluster randomized trial. Contemp Clin Trials Commun. 2022 Mar 9;27:100907. doi: 10.1016/j.conctc.2022.100907. eCollection 2022 Jun. PMID 35499065